CLINICAL TRIAL: NCT05150990
Title: Using Rendever to Improve the Quality of Life of Older Adults With Cognitive Impairments in Senior Living Communities and Their Family Members Who Live at a Distance
Brief Title: Technology and Family Thriving Study
Acronym: Thrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Collaborators: Rendever, Inc. (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nancy Collins, Professor, University of California, Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIH 13336607; R42AG063640-02 (NIH); 3R42AG063640-03S1 (NIH)
Record Dates: First submitted 2021-10-28; First posted 2021-12-09 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Dementia; Caregiver Burnout; Quality of Life; Mental Health Wellness 1; Loneliness; Family Relationship
Keywords: Virtual reality; Video chat (Zoom); Technology; Senior living community; Seniors; Older adults; Cognitive impairment; Dementia; Thriving; Quality of Life; Loneliness; Mental health; Caregiver guilt; Caregiver burden; Family relationships; Adult children; Assisted living; Social connection
MeSH Terms: conditions — Alzheimer Disease; Dementia; Caregiver Burden; Cognitive Dysfunction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Dyads (older adult and adult child) will be randomly assigned to one of two intervention groups (two types of technology): (1) virtual reality, or (2) video chat (active control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Weekly activities using virtual reality (Rendever)
  Interventions: Behavioral: Virtual Reality
- Video Chat (Active Comparator): Weekly activities using video conference (Zoom)
  Interventions: Behavioral: Video Chat

INTERVENTIONS:
Behavioral: Virtual Reality — Older adults (residents of senior living communities) engage in four 20-minute virtual reality activities (via the Rendever platform) with their adult child each week for 4 consecutive weeks. The 4 sessions include immersive virtual adventures (e.g., bucket list travel) and reminiscence activities (e.g., virtual life story). Adult children participate remotely from their own homes.
  Arms: Virtual Reality
Behavioral: Video Chat — Older adults (residents of senior living communities) engage in four 20-minute video chat sessions (via the Zoom platform) with their adult child each week for 4 consecutive weeks. Adult children participate remotely from their own homes.
  Arms: Video Chat

SUMMARY:
The purpose of this project is to test the impact of different forms of technology (virtual reality vs. video chat) on quality of life and family relationships in older adults who reside in senior living communities and an adult child who lives at a distance. The study will also investigate whether responses to the technology and quality of life outcomes depend on older adults' level of cognitive impairment.

DETAILED DESCRIPTION:
Purpose of the clinical trial: The virtual reality (VR) program, Rendever, enables older adults in senior living communities to maintain important family relationships, engage fully with life, and reconnect with their past, regardless of physical location, through its advanced networking and live-streaming capabilities. This project will test the immediate and longer-term impact of the Rendever virtual reality platform (vs. video chat) on the quality of life of residents and their adult children in an experimental design. The study will also investigate whether responses to the technology and quality of life outcomes depend on older adults' level of cognitive impairment.

Participants: Participants will be older adults (age 50+) with mild cognitive impairments (MCI) or mild to moderate Alzheimer's Disease or related dementias (ADRD) who reside in senior living communities and an adult child who lives at a distance. The resident-adult child dyads (target N=192 dyads) will be recruited from 12 senior living communities in the greater Boston area and central California. Residents will participate from their senior living community and adult children will participate from their own home, at least 45 minutes driving distance away.

Study Design and Method: The design is a 2 (Intervention Group: Virtual Reality vs. Active Control) x 2 (Level of Cognitive Impairment: MCI vs. ADRD) x Time (7 time points) design. Dyads will be randomly assigned to an intervention group (Virtual Reality vs. Video Chat Control). Dependent variables will include quality of life, psychological and social well-being (loneliness, mental health, thriving, and relationship quality), caregiver guilt (guilt, stress, and burden), and positive engagement while using the technology. Outcomes will be assessed through surveys, interviews, and observational methods.

The experimental intervention will be implemented in a between-group design. Dyads will be randomly assigned to either the Virtual Reality Condition or the active Control Condition (video chat). Participants will complete a baseline survey (T1), followed by four activity sessions once a week for 4 consecutive weeks (T2-T5). Follow-up surveys will be conducted at 1-month (T6) and 3-months (T7) post-intervention for exploratory purposes (to determine if any effects of the technology are sustained over time). Residents and adult children will also be interviewed briefly after the intervention and at each follow-up. All sessions will be video and audiotaped. Computerized and human coding will examine positive engagement and interpersonal dynamics while using the technology.

Dyads assigned to the virtual reality (VR) condition will engage in 4 weekly VR sessions that include immersive virtual adventures (e.g., bucket list travel) and reminiscence activities (e.g., virtual life story). Dyads assigned to the control condition will engage in 4 weekly video chat sessions. During these sessions, dyads will engage in conversations that are typical in their daily lives. All other procedures will be identical in the two conditions.

Sample size, recruitment, and statistical power: A power analysis using simulation methods (for multi-level regression models and structural equation models) was used to determine the sample size. A sample size of 192 dyads (96 in each intervention condition) evenly split between cognitive impairment groups (MCI vs. dementia) will achieve a high level of power for detecting the minimal expected effect size (accounting for expected attrition).

Statistical analysis: Because data from parent-adult child dyads will be dependent, and because the dyad is the unit of analysis for assignment to experimental conditions, the analysis of quantitative data will utilize linear models designed for nested (clustered) data. Hypothesis testing will be conducted with multi-level, random-effects regression and multi-level structural equation modeling.

Study Aims:

AIM 1: Determine whether virtual reality (vs. control) improves quality of life for residents and their adult children who live at a distance.

AIM 2: Determine whether the positive effects of virtual reality (vs. control) on quality of life depend upon residents' level of cognitive impairment (MCI vs. mild to moderate AD/ADRD).

AIM 3: Determine whether virtual reality (vs. control) reduces caregiver guilt for adult children and whether these effects depend on the adult child's own responses to the technology and their parent's responses to the technology.

ELIGIBILITY:
Inclusion Criteria for older adults:

* Must reside in one of the senior living communities participating in the study
* at least 50 years old
* Fluent in English or Spanish
* Have MCI or mild to moderate AD/ADRD
* Mini-mental state examination (MMSE-2) score between 13 and 27
* Have an adult child who lives at least 45 minutes driving distance from the community and is willing to participate with them
* Do not have an overly negative, aggressive, or abusive relationship with this adult child

Inclusion Criteria for adult children:

* At least 18 years old
* Fluent in English or Spanish,
* Live at least 45 minutes driving distance from the residential community
* Do not have an overly negative, aggressive, or abusive relationship with their parent

Exclusion Criteria:

* Severe AD/ADRD (MMSE-2 score < 13)
* History of seizure, severe vertigo, hallucinations, or aggression
* Severe visual impairment (screening will be conducted to determine if vision is sufficient to participate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Afifi, PhD, Principal Investigator — University of California, Santa Barbara; Kyle Rand, B.A., Principal Investigator — Rendever Co.; Nancy Collins, PhD, Principal Investigator — University of California, Santa Barbara
Locations (27):
- United States (27):
  - Belmont Calabasas, Calabasas, California
  - Oakmont of Camarillo, Camarillo, California
  - Friendship Manor, Goleta, California
  - Casa Dorinda, Montecito, California
  - Ojai Gables, Ojai, California
  - Garden Court on De La Vina, Santa Barbara, California
  - Covenant Living at the Samarkand, Santa Barbara, California
  - Gardens on Hope, Santa Barbara, California
  - Grace Village Apartments, Santa Barbara, California
  - Valle Verde, Santa Barbara, California
  - Vista Del Monte, Santa Barbara, California
  - Heritage House, Santa Barbara, California
  - Maravilla, Santa Barbara, California
  - Atterdag Village of Solvang, Solvang, California
  - Stone Hill at Andover, Andover, Massachusetts
  - Stonebridge at Burlington, Burlington, Massachusetts
  - Youville House Assisted Living, Cambridge, Massachusetts
  - Cadbury Commons, Cambridge, Massachusetts
  - Brightview Canton, Canton, Massachusetts
  - The Linden at Danvers, Danvers, Massachusetts
  - Brightview North Andover, North Andover, Massachusetts
  - Benchmark of Norwood (Clapboardtree), Norwood, Massachusetts
  - Laurelwood at The Pinehills, Plymouth, Massachusetts
  - Autumn Glen at Dartmouth, South Dartmouth, Massachusetts
  - Bayberry at Emerald Court, Tewksbury, Massachusetts
  - Carriage House at Lee's Farm, Wayland, Massachusetts
  - Ledgewood Bay Assisted Living, Milford, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data and related information will be made available to researchers and data analysts at no cost through NACDA-Open Aging Repository (NACDA-OAR), which is an NIH-funded repository. Quantitative data, codebooks, descriptions of missing data, and any errors will be made available on the site. The data submitted will conform to the NACDA-OAR standards.
Supporting Information: Study Protocol, ICF
Time Frame: Deidentified data and related files will be made available in the NACDA-OAR repository no later than within one year of the completion of the funded project period or upon the first publication of the data online. Data will be posted indefinitely.
Access Criteria: Data will be deposited and made available through NACDA-Open Aging Repository (NACDA-OAR) and will be shared with investigators working under an institution with a Federal Wide Assurance (FWA). Data can be used for secondary study purposes. Users will be required to register on the password-protected site in order to access the data files, which includes agreeing to the conditions of use related to the public release of the data. This includes not using any identifying information, ethical reporting, not selling the data to third parties, acknowledging the data source, and destroying the data upon use.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Older adults with cognitive impairment and an adult child were recruited at 23 senior living communities in two geographic regions in the U.S. (Boston, MA, and Santa Barbara, CA) between October 2021 and December 2023, with the trial's primary completion in March 2024. Approximately half the older adults had mild cognitive impairment (MCI) and half had mild to moderate Alzheimer's disease or related dementias (ADRD). A total of 186 dyads (372 participants) were enrolled.
Groups:
- Video Chat: Weekly activities using video conference (Zoom)
  Video Chat (Active Control): Older adults engage in four 20-minute video chat sessions (via the Zoom platform) with their adult child each week for 4 consecutive weeks. Adult children participate remotely from their own homes.
- Virtual Reality: Weekly activities using virtual reality (Rendever)
  Virtual Reality: Older adults engage in four 20-minute virtual reality activities (via the Rendever platform) with their adult child each week for 4 consecutive weeks. The 4 sessions include immersive virtual adventures (e.g., bucket list travel) and reminiscence activities (e.g., virtual life story). Adult children participate remotely from their own homes.
Period: Overall Study
Arm/Group | Video Chat | Virtual Reality
Started | 96 (Participant flow values refer to the number of dyads, not individuals. 96 dyads (96 older adult participants and 96 adult child participants) were randomly assigned to the "Video Chat" arm.) | 90 (Participant flow values refer to the number of dyads, not individuals. 90 dyads (90 older adult participants and 90 adult child participants) were randomly assigned to the "Virtual Reality" arm.)
Baseline Assessment | 96 (The baseline assessment included two surveys, an intake survey (demographic and health information) and a baseline survey (initial assessment of all primary outcomes). The intake survey was completed by all 96 dyads. The baseline survey was completed by at least one member of 94 dyads (94 older adults and 93 adult children) in the "Video Chat" arm.) | 90 (The baseline assessment included two surveys, an intake survey (demographic and health information) and a baseline survey (initial assessment of all primary outcomes). The intake survey was completed by all 90 dyads. The baseline survey was completed by at least one member of 88 dyads (87 older adults and 88 adult children) in the "Virtual Reality" arm.)
Started Intervention | 92 (The intervention was started by 92 dyads (92 older adults and 92 adult children) in the "Video Chat" arm.) | 84 (The intervention was started by 84 dyads (84 older adults and 84 adult children) in the "Virtual Reality" arm.)
Completed Intervention | 87 (The intervention was completed by 87 dyads (87 older adults and 87 adult children) in the "Video Chat" arm.) | 79 (The intervention was completed by 79 dyads (79 older adults and 79 adult children) in the "Virtual Reality" arm.)
Completed Post-Intervention Assessment | 87 (The post-intervention assessment was completed by at least one member of 87 dyads (87 older adults and 86 adult children) in the "Video Chat" arm.) | 79 (The post-intervention assessment was completed by at least one member of 79 dyads (79 older adults and 78 adult children) in the "Virtual Reality" arm.)
1-Month Follow-up Assessment | 86 (The 1-month assessment was completed by at least one member of 86 dyads (86 older adults and 85 adult children) in the "Video Chat" arm.) | 79 (The 1-month assessment was completed by at least one member of 79 dyads (79 older adults and 78 adult children) in the "Virtual Reality" arm.)
3-Month Follow-Assessment | 84 (The 3-month assessment was completed by at least one member of 84 dyads (84 older adults and 84 adult children) in the "Video Chat" arm.) | 78 (The 3-month assessment was completed by at least one member of 78 dyads (78 older adults and 77 adult children) in the "Virtual Reality" arm.)
Completed | 84 (The study was completed by at least one member of 84 dyads (84 older adults and 84 adult children) in the "Video Chat" arm.) | 78 (The study was completed by at least one member of 78 dyads (78 older adults and 77 adult children) in the "Virtual Reality" arm.)
Not Completed | 12 | 12
Not completed — Decline in health of older adult (unrelated to the intervention) | 5 | 2
Not completed — Dissatisfaction with surveys (length, time commitment, too personal) or other study procedures | 6 | 2
Not completed — Adverse response to the intervention - social strain | 0 | 2
Not completed — Adverse response to the intervention - discomfort using technology | 0 | 1
Not completed — External circumstances (family emergency, loss of Wifi) | 0 | 2
Not completed — Participant no longer eligible due to history of seizures not previously reported | 0 | 1
Not completed — Death (unrelated to the intervention) | 1 | 2

BASELINE CHARACTERISTICS:
Population: A total of 186 dyads (372 individuals) enrolled and completed a brief intake survey on demographics and health. Of these, 96 dyads (N=193) were assigned to the Video Chat arm and 90 (N=180) to the Virtual Reality arm. The intake survey was completed at enrollment; the full baseline survey occurred later, after some dyads withdrew. Thus, the number of baseline cases may vary slightly depending on the source of the variable being reported (intake vs. full baseline survey).
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Chat | Virtual Reality | Total
Number analyzed (Participants) | 192 | 180 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 186 dyads completed demographic information in the "intake" survey (186 older adults and 186 adult children).
  years
    Older Adults: number analyzed (Participants) | 96 | 90 | 186
    Older Adults | 85.86 (6.98) | 85.68 (8.06) | 85.77 (7.50)
    Adult Children: number analyzed (Participants) | 96 | 90 | 186
    Adult Children | 56.72 (9.63) | 56.03 (10.47) | 56.38 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 186 dyads completed demographic information in the "intake" survey (186 older adults and 186 adult children).
  Participants
    Older Adults: number analyzed (Participants) | 96 | 90 | 186
    Older Adults: Female | 67 | 61 | 128
    Older Adults: Male | 29 | 29 | 58
    Adult Children: number analyzed (Participants) | 96 | 90 | 186
    Adult Children: Female | 61 | 50 | 111
    Adult Children: Male | 35 | 40 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 186 dyads completed demographic information in the "intake" survey (186 older adults and 186 adult children).
  Participants
    Older Adults: number analyzed (Participants) | 96 | 90 | 186
    Older Adults: Hispanic or Latino | 2 | 5 | 7
    Older Adults: Not Hispanic or Latino | 93 | 85 | 178
    Older Adults: Unknown or Not Reported | 1 | 0 | 1
    Adult Children: number analyzed (Participants) | 96 | 90 | 186
    Adult Children: Hispanic or Latino | 2 | 5 | 7
    Adult Children: Not Hispanic or Latino | 94 | 84 | 178
    Adult Children: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 186 dyads completed demographic information in the "intake" survey (186 older adults and 186 adult children).
  Participants
    Older Adults: number analyzed (Participants) | 96 | 90 | 186
    Older Adults: American Indian or Alaska Native | 0 | 0 | 0
    Older Adults: Asian | 0 | 1 | 1
    Older Adults: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Older Adults: Black or African American | 1 | 0 | 1
    Older Adults: White | 94 | 87 | 181
    Older Adults: More than one race | 0 | 2 | 2
    Older Adults: Unknown or Not Reported | 1 | 0 | 1
    Adult Children: number analyzed (Participants) | 96 | 90 | 186
    Adult Children: American Indian or Alaska Native | 0 | 0 | 0
    Adult Children: Asian | 2 | 1 | 3
    Adult Children: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Adult Children: Black or African American | 1 | 0 | 1
    Adult Children: White | 90 | 87 | 177
    Adult Children: More than one race | 1 | 1 | 2
    Adult Children: Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants] — This table shows the region of enrollment for all individuals in the study (rather than dyads) because dyad members did not necessarily reside in the same location. All older adults were enrolled and participated in the U.S.; eight adult children participated remotely from outside the U.S.
  participants
    United States | 189 | 175 | 364
    Australia | 0 | 1 | 1
    Canada | 1 | 0 | 1
    Colombia | 0 | 1 | 1
    Denmark | 0 | 1 | 1
    Germany | 1 | 1 | 2
    Saudi Arabia | 1 | 0 | 1
    Switzerland | 0 | 1 | 1
Cognitive Group (MCI/ADRD) - Older adults [Count of Participants; unit: Participants] — Level of cognitive impairment was assessed only for older adult participants (not for adult children). MCI = Mild cognitive impairment. ADRD = mild to moderate Alzheimer's disease or related dementia. Population: Cognitive group (MCI/ADRD) was assessed only for the older adult member of each dyad.
  Participants
    number analyzed (Participants) | 96 | 90 | 186
    MCI | 44 | 41 | 85
    ADRD | 52 | 49 | 101

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life in Alzheimer's Disease (QOL-AD) - Changes From Baseline (Older Adult)
Description: QOL-AD (R.G. Logsdon, 1996) is a 13-item self-report measure of quality of life (completed by older adult participants). (As a secondary outcome, adult children also reported on their parents' quality of life). Items are rated on a 4-point scale: 1 = Poor, 2 = Fair, 3 = Good, 4 = Excellent. The total score is the mean of all items (range: 1 to 4). Higher scores indicate greater quality of life.
Time Frame: T1 (baseline, 1-week pre-intervention), T2 (1-week post-intervention), T3 (1-month post-intervention), T4 (3-months post-intervention)
Population: Some participants withdrew from the study after the T1 (baseline) assessment. Several others remained in the study but failed to complete the T2 (post-intervention) assessment. Primary aims focus on changes from T1 (Baseline) to T2 (1-week Post-Intervention). T3 and T4 are exploratory and not presented here.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MCI Group/Video Chat: Tech Condition = Video Chat (Zoom) Cognitive group = Older adults with mild cognitive impairment (MCI)
- MCI Group/Virtual Reality: Tech Condition = Virtual Reality (Rendever) Cognitive Group = Older adults with mild cognitive impairment (MCI)
- ADRD Group/Video Chat: Tech Condition = Video Chat (Zoom) Cognitive group = Older adults with mild to moderate Alzheimer's disease or related dementia (ADRD)
- ADRD Group/Virtual Reality: Tech Condition = Virtual Reality (Rendever) Cognitive Group = Older adults with mild to moderate Alzheimer's disease or related dementia (ADRD)
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 48
score on a scale
  T1 (Baseline) | 3.04 (0.41) | 3.00 (0.48) | 2.85 (0.49) | 2.94 (0.44)
  T2 (Post-Intervention): number analyzed (Participants) | 41 | 38 | 45 | 40
  T2 (Post-Intervention) | 3.08 (0.36) | 2.98 (0.51) | 2.91 (0.44) | 3.07 (0.38)

2. Primary Outcome: Brief Inventory of Thriving (BIT) - Changes From Baseline (Older Adult)
Description: An 11-item measure of thriving adapted from the Brief Inventory of Thriving (BIT) and the Comprehensive Inventory of Thriving (CIT; Su, R., Tay, L., & Diener, E., 2014). This measure provides a holistic view of positive functioning (completed by older adults and adult children). Items are rated on a 5-point scale: 1 = Strongly Disagree, 2 = Disagree, 3 = Neither Agree nor Disagree, 4 = Agree, 5 = Strongly Agree. The total score is the average of the 11 items (range: 1 to 5). Higher scores indicate a greater sense of thriving.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 48 | 47
score on a scale
  T1 - Older Adult | 3.97 (0.59) | 3.90 (0.58) | 3.63 (0.65) | 3.69 (0.56)
  T2 - Older Adult: number analyzed (Participants) | 41 | 38 | 45 | 40
  T2 - Older Adult | 4.00 (0.53) | 3.89 (0.68) | 3.62 (0.64) | 3.91 (0.52)

3. Primary Outcome: Positive and Negative Affect Schedule (PANAS) - Changes From Baseline (Older Adult)
Description: This scale includes 12 items from the longer PANAS (Watson, Clark, & Tellegen, 1988), which measures two primary dimensions of mood. (Completed by older adults and adult children.) Participants rate the extent to which they experienced positive and negative emotions over the past week. Each item is rated on a 5-point scale: 1 = Not at all, 2 = A little, 3 = Moderately, 4 = Quite a lot, 5 = Extremely. Separate subscale scores are calculated for positive emotion (6 items) and negative emotion (6 items) by averaging responses within each set (range: 1 to 5). Higher scores on the positive emotion subscale reflect greater positive mood during the past week, indicating better well-being. Higher scores on the negative emotion subscale reflect greater negative mood, indicating poorer well-being.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 48
score on a scale
  T1 - Positive Emotions | 3.72 (0.68) | 3.73 (0.72) | 3.20 (0.91) | 3.18 (0.84)
  T2 - Positive Emotions: number analyzed (Participants) | 41 | 38 | 45 | 39
  T2 - Positive Emotions | 3.76 (0.58) | 3.65 (0.63) | 3.33 (0.87) | 3.53 (0.60)
  T1 - Negative Emotions | 1.74 (0.51) | 1.90 (0.75) | 1.96 (0.82) | 1.65 (0.58)
  T2 - Negative Emotions: number analyzed (Participants) | 41 | 38 | 45 | 39
  T2 - Negative Emotions | 1.46 (0.42) | 1.70 (0.61) | 1.71 (0.64) | 1.54 (0.74)

4. Primary Outcome: Geriatric Depression Scale (GDS) - Changes From Baseline (Older Adult)
Description: GDS (Sheikh, J.I., & Yesavage, J.A., 1986) is a 15-item self-report measure of depression (completed by older adult participants). Items are rated "Yes" or "No" and are scored "1" if the response reflects depressive symptoms. Total score is the sum of all items (range: 0 to 15). Higher scores indicate greater depression.
Time Frame: as for outcome 1
Population: Some participants withdrew from the study after the T1 (baseline) assessment or remained in the study but failed to complete the T2 (post-intervention) assessment. Primary aims focus on changes from T1 (Baseline) to T2 (1-week Post-Intervention). T3 and T4 are exploratory and not presented here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 48
score on a scale
  T1 (Baseline) | 1.95 (2.16) | 2.73 (2.74) | 3.20 (2.98) | 2.82 (1.79)
  T2 (Post-Intervention): number analyzed (Participants) | 41 | 38 | 45 | 40
  T2 (Post-Intervention) | 1.81 (2.16) | 3.20 (3.39) | 3.35 (2.99) | 2.34 (1.79)

5. Primary Outcome: Mental Health Inventory (MHI) - Changes From Baseline (Older Adult)
Description: The MHI includes 5 items from the longer MHI (McHorney, Ware, & Raczek, 1993) to assess depression, anxiety, and vitality during the past week (completed by older adults and adult children). Items are rated on a 6-point scale: 1= None of the time, 2= A little of the time, 3 = Some of the time, 4 = A good bit of the time, 5 = Most of the time, 6 = All of the time. The total score is the average of all 8 items, some reverse-scored (range: 1 to 6). Higher scores indicate better mental health.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 48
score on a scale
  T1 (Baseline) | 5.22 (0.52) | 4.88 (0.87) | 4.81 (0.81) | 5.06 (.66)
  T2 (Post-Intervention): number analyzed (Participants) | 41 | 38 | 43 | 40
  T2 (Post-Intervention) | 5.19 (0.61) | 5.08 (0.74) | 4.94 (0.75) | 5.05 (0.72)

6. Primary Outcome: Revised UCLA Loneliness Scale (Short Form) - Changes From Baseline (Older Adult)
Description: The short form of the Revised UCLA Loneliness Scale (Hughes, Waite, Hawkley, & Cacioppo, 2008) is a 4-item scale widely used in field research with older adults, and adapted from the original scale (Russell D, Peplau LA, Cutrona CE, 1980). Items are rated on a 4-point scale: 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often. The total score is the mean of the 4 items (range: 1 to 4). Higher scores indicate greater loneliness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 48
score on a scale
  T1 (Baseline) | 1.98 (0.75) | 1.86 (0.81) | 1.96 (.073) | 1.81 (0.67)
  T2 (Post-Intervention): number analyzed (Participants) | 41 | 38 | 49 | 48
  T2 (Post-Intervention) | 1.71 (0.67) | 1.73 (0.79) | 1.95 (0.83) | 1.86 (0.87)

7. Primary Outcome: Unidimensional Relationship Closeness Scale - Changes From Baseline (Older Adult)
Description: Relationship closeness is assessed with 4 items from the Unidimensional Relationship Closeness Scale (Dibble, Levine, & Park, 2011). (Completed by older adults and adult children). Items are rated on a 7-point scale: 1 = Strongly disagree, 2 = Disagree, 3 = Somewhat disagree, 4 = Neutral, 5 = Somewhat agree, 6 = Agree, 7 = Strong Agree. The total score is the average of the 4 items (range: 1 to 7). Higher scores indicate greater relationship closeness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 48
score on a scale
  T1 - Older Adult | 5.94 (1.11) | 6.29 (0.65) | 6.07 (0.75) | 5.78 (1.25)
  T2 - Older Adult: number analyzed (Participants) | 41 | 38 | 45 | 40
  T2 - Older Adult | 6.28 (0.74) | 6.39 (0.60) | 6.22 (0.72) | 6.18 (1.01)

8. Primary Outcome: Relationship Satisfaction - Changes From Baseline (Older Adult)
Description: Global relationship satisfaction is assessed with 3 items adapted from Huston et al.'s (1986) relationship satisfaction scale (completed by older adults and adult children). Items are rated on a 6-point scale: 1 = Not at all, 2 = A little, 3 = Somewhat, 4 = Very, 5 = Almost completely, 6 = Completely. Total scores are the average of the 3 items (range: 1 to 6). Higher scores indicate greater relationship satisfaction.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 48 | 47
score on a scale
  T1 - Older Adult | 4.92 (1.21) | 5.17 (1.06) | 4.88 (1.17) | 4.99 (1.17)
  T2 - Older Adult: number analyzed (Participants) | 41 | 38 | 45 | 40
  T2 - Older Adult | 5.11 (0.95) | 4.24 (0.87) | 5.07 (0.95) | 5.19 (1.18)

9. Primary Outcome: Communal Coping - Changes From Baseline (Older Adult)
Description: Communal coping is assessed with 3 items reflecting feelings of unity when combatting stress (Afifi et al., 2019). (Completed by older adults and adult children.) Items are rated on a 5-point scale: 1 = Strongly disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, 5 = Strongly agree. The total score is the average of the 3 items (range: 1 to 5). Higher scores indicate a greater sense of communal coping.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 39 | 49 | 46
score on a scale
  T1 - Older Adult | 3.91 (0.77) | 3.94 (0.78) | 3.89 (0.85) | 3.93 (0.82)
  T2 - Older Adult: number analyzed (Participants) | 41 | 38 | 45 | 40
  T2 - Older Adult | 3.99 (0.77) | 3.98 (0.67) | 3.99 (0.71) | 4.14 (0.80)

10. Primary Outcome: Brief Inventory of Thriving (BIT) - Changes From Baseline (Adult Child)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 50 | 47
score on a scale
  T1 - Adult Child | 4.04 (0.54) | 4.22 (0.42) | 4.15 (0.51) | 4.02 (0.55)
  T2 - Adult Child: number analyzed (Participants) | 39 | 37 | 44 | 40
  T2 - Adult Child | 4.18 (0.50) | 4.31 (0.33) | 4.11 (0.54) | 4.09 (0.44)

11. Primary Outcome: Center for Epidemiological Studies Depression Scale Revised Short Form (CESD-R-10) - Changes From Baseline (Adult Child)
Description: The CESD-R-10 (Björgvinsson, Kertz, Bigda-Peyton, McCoy, Aderka,2013) is a 10-item measure of depressive symptoms adapted from the longer CESD (completed by adult children). Participants are asked to report how they felt during the past week. Items are rated on a 4-point scale: 0 = Rarely or none of the time, 1 = Some or a little of the time, 2 = Occasionally or a moderate amount of the time, 3 = Most or all of the time. The total score is the mean of the 10 items, some reverse-scored (range: 0 to 3). Higher scores reflect more depressive symptoms, worse mental health.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 47
score on a scale
  T1 (Baseline) | 0.57 (0.42) | 0.42 (0.29) | .48 (0.48) | 0.53 (0.44)
  T2 (Post-Intervention): number analyzed (Participants) | 39 | 37 | 44 | 40
  T2 (Post-Intervention) | 0.48 (0.44) | 0.33 (0.27) | 0.49 (0.45) | 0.47 (0.46)

12. Primary Outcome: Positive and Negative Affect Schedule (PANAS) - Changes From Baseline (Adult Child)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 50 | 48
score on a scale
  T1 - Positive Emotions | 3.99 (0.72) | 3.75 (0.53) | 3.56 (0.63) | 3.58 (0.53)
  T2 - Positive Emotions: number analyzed (Participants) | 39 | 36 | 44 | 40
  T2 - Positive Emotions | 3.51 (0.65) | 3.89 (0.45) | 3.59 (0.62) | 3.67 (0.55)
  T1 - Negative Emotions | 1.73 (0.45) | 1.70 (0.36) | 1.78 (0.56) | 1.73 (0.46)
  T2 - Negative Emotions: number analyzed (Participants) | 39 | 36 | 44 | 40
  T2 - Negative Emotions | 1.64 (0.56) | 1.53 (0.35) | 1.77 (0.61) | 1.59 (0.43)

13. Primary Outcome: Mental Health Inventory (MHI) - Changes From Baseline (Adult Child)
Description: The MHI includes 5 items from the longer MHI (McHorney, Ware, & Raczek, 1993) to assess depression, anxiety, and vitality during the past week (completed by older adults and adult children). Items are rated on a 6-point scale: 1 = None of the time, 2 = A little of the time, 3 = Some of the time, 4 = A good bit of the time, 5 = Most of the time, 6 = All of the time. The total score is the average of all 8 items, some reverse-scored (range: 1 to 6). Higher scores indicate better mental health.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 50 | 47
score on a scale
  T1 (Baseline) | 4.88 (0.68) | 5.05 (0.54) | 4.98 (0.62) | 4.95 (0.63)
  T2 (Post-Intervention): number analyzed (Participants) | 39 | 36 | 46 | 41
  T2 (Post-Intervention) | 4.96 (0.77) | 5.02 (0.76) | 5.03 (0.71) | 5.18 (0.58)

14. Primary Outcome: Perceived Stress Scale (PSS) - Changes From Baseline (Adult Child)
Description: The PSS short form (completed by adult children) is a 4-item scale adapted from the longer PSS (Cohen, Kamarck, & Mermelstein, 1983). Items are rated on a 5-point scale: 1 = Never, 2 = Almost never, 3 = Sometimes, 4 = Fairly often, 5 = Very often. The total score is the average of the 4 items, some reverse-scored (range: 1 to 5). Higher scores indicate greater perceived stress.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 50 | 47
score on a scale
  T1 - Baseline | 2.13 (0.65) | 1.89 (0.54) | 2.17 (0.64) | 2.02 (0.64)
  T2 - Post-Intervention: number analyzed (Participants) | 39 | 36 | 45 | 41
  T2 - Post-Intervention | 1.97 (.60) | 1.89 (0.71) | 1.99 (0.69) | 1.83 (0.69)

15. Primary Outcome: Caregiver Guilt/Grief Scale - Changes From Baseline (Adult Child)
Description: This scale (completed by adult children) includes 13 items adapted from the caregiver guilt and grief scales (Wells, Jorm, Jordan, & Lefroy, 1990). Items are rated on a 5-point scale: 1= Not at all, 2 = A little, 3 = A moderate amount, 4 = A lot, 5 = Almost unbearably. The total score is the average of the 13 items (range: 1 to 5). Higher scores indicate greater caregiver guilt/grief.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 47
score on a scale
  T1 (Baseline) | 1.77 (0.45) | 2.00 (0.66) | 2.15 (0.69) | 1.99 (0.72)
  T2 (Post-Intervention): number analyzed (Participants) | 39 | 37 | 44 | 40
  T2 (Post-Intervention) | 1.74 (0.48) | 1.99 (0.63) | 2.12 (0.75) | 2.06 (0.64)

16. Primary Outcome: Relational Burnout/Load Scale - Changes From Baseline (Adult Child)
Description: Relational burnout/load is assessed with 6 items from the Relational Load Scale (Afifi et al., 2019). (Completed by adult children.) Items are rated on a 5-point scale: 1 = Strongly disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, 5 = Strongly agree. The total score is the average of the 6 items, some reverse-scored (range: 1 to 5). Higher scores indicate a greater sense of relational load/burnout.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 47
score on a scale
  T1 (Baseline) | 1.80 (0.68) | 1.82 (0.57) | 1.95 (0.70) | 1.89 (0.72)
  T2 (Post-Intervention) | 1.76 (0.58) | 1.87 (0.64) | 1.88 (0.66) | 1.90 (0.72)

17. Primary Outcome: Unidimensional Relationship Closeness Scale - Changes From Baseline (Adult Child)
Description: Relationship closeness is assessed with 4 items from the Unidimensional Relationship Closeness Scale (Dibble, Levine, & Park, 2011). (Completed by older adults and adult children.) Items are rated on a 7-point scale: 1 = Strongly disagree, 2 = Disagree, 3 = Somewhat disagree, 4 = Neutral, 5 = Somewhat agree, 6 = Agree, 7 = Strong Agree. The total score is the average of the 4 items (range: 1 to 7). Higher scores indicate greater relationship closeness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 47
score on a scale
  T1 (Baseline) | 5.36 (1.53) | 5.80 (1.01) | 5.58 (1.13) | 5.67 (1.08)
  T2 (Post-Intervention): number analyzed (Participants) | 39 | 37 | 44 | 40
  T2 (Post-Intervention) | 5.84 (1.31) | 5.78 (1.07) | 5.65 (1.15) | 5.44 (1.25)

18. Primary Outcome: Relationship Satisfaction - Changes From Baseline (Adult Child)
Description: Global relationship satisfaction is assessed with 3 items adapted from Huston et al.'s (1986) relationship satisfaction scale (completed by older adults and adult children). Items are rated on a 6-point scale: 1 = Not at all, 2 = A little, 3 = Somewhat, 4 = Very, 5 = Almost completely, 6 = Completely. The total score is the average of the 3 items (range: 1 to 6). Higher scores indicate greater relationship satisfaction.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 47
score on a scale
  T1 (Baseline) | 4.38 (1.21) | 4.35 (1.29) | 4.08 (1.16) | 4.17 (1.27)
  T2 (Post-Intervention): number analyzed (Participants) | 39 | 37 | 44 | 40
  T2 (Post-Intervention) | 4.70 (0.99) | 4.41 (1.26) | 4.21 (1.17) | 4.32 (1.23)

19. Primary Outcome: Communal Coping - Changes From Baseline (Adult Child)
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCI Group/Video Chat | MCI Group/Virtual Reality | ADRD Group/Video Chat | ADRD Group/Virtual Reality
Number analyzed (Participants) | 43 | 40 | 49 | 47
score on a scale
  T1 (Baseline) | 3.31 (0.98) | 3.39 (0.87) | 3.24 (0.83) | 3.12 (1.09)
  T2 (Post-Intervention): number analyzed (Participants) | 39 | 37 | 44 | 40
  T2 (Post-Intervention) | 3.56 (0.93) | 3.46 (0.98) | 3.34 (0.79) | 3.32 (1.03)

20. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) - Technology Sessions
Description: Positive and negative emotions experienced during the technology session (older adult and adult child). Rated on a scale from 1 to 5, and separate indexes are computed for positive emotion and negative emotion. Higher scores represent greater positive and negative emotion. Scores will be averaged across the intervention period (4 weeks) for overall measures of positive/negative affect experienced during the intervention. Higher positive emotion and lower negative emotion indicate a more favorable response during the technology session.
Time Frame: Immediately after each of the 4 technology sessions during the intervention (one week apart)
Reporting Status: Not Posted, anticipated posting 2025-09

21. Secondary Outcome: Social and Conversational Engagement - Technology Sessions
Description: Social and conversational engagement during the technology sessions will be evaluated using items developed specifically for this study, based on findings from a pilot study. Higher scores indicate greater engagement. Engagement scores will be averaged over the four-week intervention period to generate an overall engagement measure. In addition to self-reports, objective coders will analyze video and audio recordings of the sessions to assess conversational and emotional engagement. Kinesic (physical) engagement of the older adult will be evaluated both by trained raters and an automated computer program.
Time Frame: Immediately after each of the 4 technology sessions during the intervention (one week apart)
Reporting Status: Not Posted, anticipated posting 2025-09

22. Secondary Outcome: Relationship Satisfaction and Communication Quality - Technology Sessions
Description: Multiple items designed to assess features of relationship quality (older adult and adult child). Higher scores represent greater satisfaction and communication quality. Scores will be averaged across the intervention period (4 weeks) for an overall score of relationship satisfaction and communication quality during the technology sessions, during the intervention period.
Time Frame: Immediately after each of the 4 technology sessions during the intervention (one week apart)
Reporting Status: Not Posted, anticipated posting 2025-09

23. Secondary Outcome: Telepresence and Copresence - Technology Session
Description: Rating of engagement and immersion during the technology session (older adult and adult child). Items were written for this project based on a pilot study. Higher scores represent greater telepresence and co-presence. Due to time limitations, this measure is completed only during the first technology session.
Time Frame: Measured after the first technology session (Week 1 of the intervention)
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: 4 months (participant enrollment through 3-month follow-up)
Description: All-Cause Mortality, Serious Adverse Events, and Other Adverse Events were reported for older adult participants. All-cause Mortality, Serious Adverse Events, and Other Adverse Events were not monitored/assessed in adult child participants.
Groups:
- Video Chat: Weekly activities using video conference (Zoom)
  Video Chat (Active Control): Older adults (residents of senior living communities) engage in four 20-minute video chat sessions (via the Zoom platform) with their adult child each week for 4 consecutive weeks. Adult children participate remotely from their own homes.
Arm/Group | Video Chat | Virtual Reality
All-Cause Mortality (participants affected / at risk) | 2/96 | 2/90
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/90
Other Adverse Events (participants affected / at risk) | 3/96 | 2/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video Chat (N=96) | Virtual Reality (N=90)
Hospitalization (General disorders) | 3 (3) | 2 (2) — Hospitalization due to unspecified illness or fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2025-03-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT05150990/Prot_SAP_006.pdf
  • Informed Consent Form: Informed Consent for Older Adult (Resident) (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05150990/ICF_007.pdf
  • Informed Consent Form: Informed Consent for Adult Child (Family Member) (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05150990/ICF_008.pdf
  • Informed Consent Form: Informed Consent for Legal Representative (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05150990/ICF_009.pdf